CLINICAL TRIAL: NCT01154140
Title: Phase 3, Randomized, Open-label Study Of The Efficacy And Safety Of Crizotinib Versus Pemetrexed/Cisplatin Or Pemetrexed/Carboplatin In Previously Untreated Patients With Non-squamous Carcinoma Of The Lung Harboring A Translocation Or Inversion Event Involving The Anaplastic Lymphoma Kinase (Alk) Gene Locus.
Brief Title: A Clinical Trial Testing The Efficacy Of Crizotinib Versus Standard Chemotherapy Pemetrexed Plus Cisplatin Or Carboplatin In Patients With ALK Positive Non Squamous Cancer Of The Lung
Acronym: PROFILE 1014
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081014; 2010-021336-33 (EudraCT Number); XALCORI (Other: Alias Study Number)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Non Squamous Lung Cancer
Keywords: open label; randomized Phase 3; first line treatment; non squamous lung cancer; ALK translocation event positive
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: treatment
- B (Active Comparator)
  Interventions: Drug: treatment

INTERVENTIONS:
Drug: treatment — crizotinib 250mg orally continuous twice daily dosing
  Arms: A
Drug: treatment — pemetrexed 500mg/m2 IV day 1 plus cisplatin 75mg/m2 IV day 1 every 21 days OR pemetrexed 500mg/m2 IV day 1 plus carboplatin AUC 5 or 6 day 1 every 21 days investigator's choice
  Arms: B

SUMMARY:
This study will evaluate the anti-cancer effects of crizotinib when compared with standard chemotherapy in patients with ALK positive lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of locally advanced not suitable for local treatment, recurrent and metastatic non-squamous cell carcinoma of the lung
* Positive for translocation or inversion events involving the ALK gene locus
* No prior systemic treatment for locally advanced or metastatic disease; Patients with brain metastases only if treated and neurologically stable with no ongoing requirement for corticosteroids
* Evidence of a personally signed and dated informed consent document and willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures including completion of patient reported outcome [PRO] measures.
* 18 years of age or older with the exception of India which has an upper age limit of 65 years old

Exclusion Criteria:

* Current treatment on another therapeutic clinical trial.
* Prior therapy directly targeting ALK.
* Any of the following within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack. - - Appropriate treatment with anticoagulants is permitted.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, uncontrolled atrial fibrillation of any grade, or QTc interval >470 msec.
* Pregnancy or breastfeeding.
* Use of drugs or foods that are known potent CYP3A4 inducers/inhibitors Concurrent use of drugs that are CYP3A4 substrates with narrow therapeutic indices.
* Known HIV infection
* Known interstitial lung disease or interstitial fibrosis
* Other severe acute or chronic medical conditions (including severe gastrointestinal conditions such as diarrhea or ulcer) or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, and which would, therefore, make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2011-01-13 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (243):
- United States (80):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - CCTAP, Fontana, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Loma Linda University Cancer Center (LLUCC)-Schuman Pavilion, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - CCTAP, Los Angeles, California
  - Kaiser Permanente Southern California, San Diego, California
  - CCTAP, San Diego, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Research Pharmacy, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lynn Cancer Institute Center for Hematology Oncology, Boca Raton, Florida
  - Florida Hospital, Orlando, Florida
  - Cancer Institute of Florida, Orlando, Florida
  - Investigational Drug Services, Orlando, Florida
  - Georgia Cancer Specialists, Athens, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Georgia Cancer Specialists, Decatur, Georgia
  - Georgia Cancer Specialists, Macon, Georgia
  - Georgia Cancer Specialists, Marietta, Georgia
  - Georgia Cancer Specialists, Sandy Springs, Georgia
  - University of Chicago, Chicago, Illinois
  - Al Fisher, Pharm D., Harvey, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Monroe Medical Associates, Harvey, Illinois
  - Monroe Medical Associates, Tinley Park, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Lois and Eskenazi Hospital, Indianapolis, Indiana
  - Monroe Medical Association, Munster, Indiana
  - The Community Hospital, Munster, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Center for Cancer Medicine, Biddeford, Maine
  - Maine Center for Cancer Medicine, Brunswick, Maine
  - Maine Center for Cancer Medicine, Sanford, Maine
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Kresge Eye Institute, Bingham Farms, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Karmanos Cancer Institute at Farmington Hills, Farmington Hills, Michigan
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Center for Advanced Medicine Infusion Center Pharmacy, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hematology-Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - UNM Eye Clinic, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - NSLIJ Health System/Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - OHSU Knight Cancer Institute, Beaverton, Oregon
  - OHSU Knight Cancer Institute, Gresham, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - OHSU Knight Cancer Institute, Tualatin, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vincent Armenio, East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt Oncology Pharmacy, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - UT Southwestern Medical Center - Simmons Cancer Center Pharmacy, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern University Hospital - William P. Clements, Jr., Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (10):
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - The Townsville Hospital, Douglas, Queensland
  - The Royal Brisbane & Womens Hospital, Herston, Queensland
  - Parkhaven Medical Center, Hyde Park, Queensland
  - Department of Medical Oncology, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Department of Haematology and Medical Oncology, East Melbourne, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
- Klinikum Wels-Grieskirchen, Wels, Austria
- Belgium (8):
  - UZ Antwerpen-Pneumologie, Edegem, Antwerp
  - Grand Hopital de Charleroi -Site Notre Dame, Charleroi, Hainaut
  - Institut Jules Bordet, Centre des Tumeurs de l'ULB, Brussels
  - Universitair Ziekenhuis Brussel / Medische Oncologie, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gent (U.Z. Gent), Ghent
  - Centre Hospitalier Universitaire de Liege, Liège
  - Department of Pulmonary Diseases AZ Delta, Roeselare
- Brazil (5):
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira - ICESP, São Paulo, São Paulo
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - R.S. McLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre (MUHC), Glen Site, Cedars Cancer Centre, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Quebec (IUCPQ), Ste-Foy, Quebec
- Chile (3):
  - Instituto Clinico Oncologico del Sur, Temuco, Cautin
  - Instituto Nacional del Cancer, Santiago, RM
  - Hospital Clinico Universidad de Chile, Seccion de Oncologia, Independencia, Santiago, Rm
- China (9):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Oncology Center, Guangdong General Hospital, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - No.81 Hospital of the PLA, Nanjing, Jiangsu
  - Oncology Department, West China Hospital of Sichuan University, Chengdu, Sichuan
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Shanghai Chest Hospital/Department of Pulmonary Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Pulmonary Hospital/Dept. of Oncology, Shanghai
- Finland (3):
  - Helsingin yliopistollinen keskussairaala, Meilahden kolmiosairaala,Keuhkosairauksien poliklinikka, Helsinki
  - Satakunnan keskussairaala/Keuhkosairauksien osasto A4, Pori
  - Tampereen yliopistollinen sairaala, Tampere
- France (9):
  - Hopital Avicenne, Bobigny
  - CHU de Caen, Caen
  - CHU Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - APHM - Hopital Nord / Service d'Oncologie Multidisciplinaire et Innovations Thérapeutiques, Marseille
  - Hopital Arnaud de Villeneuve / CHU de Montpellier, Montpellier
  - Hopital Tenon, Service de Pneumologie, Paris
  - Nouvel Hopital Civil - HSU - Pôle de Pathologie Thoracique - Service de Pneumologie, Strasbourg
- Germany (8):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Thoraxklinik am Universitaetsklinikum Heidelberg, Heidelberg
  - St.Vincentius-Kliniken Karlsruhe, Karlsruhe
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Pius-Hospital Oldenburg, Oldenburg
  - HSK Dr.- Horst-Schmidt-Kliniken GmbH,, Wiesbaden
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Department of Clinical Oncology, Queen Elizabeth Hospital, Kowloon
- India (2):
  - The Gujarat Cancer & Research Institute (M.P Shah Cancer Hospital),, Ahmedabad, Gujarat
  - Tata Memorial Centre, Tata Memorial Hospital,, Mumbai, Maharashtra
- Ireland (2):
  - Aseptic Compounding Unit, Dublin
  - Department of Medical Oncology, Dublin
- Italy (24):
  - Struttura Operativa Complessa Oncologia Medica A Centro di Riferimento Oncologico, Aviano, Pordenone
  - Farmacia, Aviano (PN)
  - Istituto dei tumori Giovanni Paolo II, Bari
  - Unità Operativa di Oncologia Medica Azienda USL Città di Bologna, Bologna
  - Azienda Ospedaliero-Universitaria "Mater Domini", Catanzaro
  - Unità Operativa di Farmacia - Campus Salvatore venuta, Catanzaro
  - Ospedale Civile Azienda USL Toscana Nord Ovest, Livorno
  - Unità Operativa Farmacia Ospedaliera PO di Livorno, Livorno
  - Fondazione IRCCS Istituto Nazionale Tumori, Struttura Complessa di Medicina Oncologica 1, Milan
  - Farmacia Istituto Europeo di Oncologia IRCCS, U.O. Farmacia, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Niguarda Ca'Granda, Divisione Oncologia Medica Falck, Milan
  - A.O.R.N. Ospedale Dei Colli - Monaldi, Napoli
  - Farmacia, Napoli
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano (TO)
  - S.C. Farmacia Ospedaliera , Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano (TO)
  - Oncologia Medica, Azienda Ospedaliero- Universitaria di Parma, Parma
  - Farmacia Ospedaliera, Perugia
  - SC Oncologia Medica, Ospedale Santa Maria della Misericordia, Perugia
  - IRCCS -Arcispedale S. Maria Nuova Tecnologie Avanzate e Modelli Assistenziali in Oncologia, Reggio Emilia
  - Istituto Regina Elena, Struttura Complessa Oncologia Medica A, Roma
  - Azienda Ospedaliera San Camillo Forlanini-Padiglione Flaiani, Roma
  - Farmacia Interna, Roma
  - Unita Operativa, Oncologia Medica, Istituto di Medicina Interna e Geriatria, Roma
- Japan (15):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kinki University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube-shi, Yamaguchi
  - National Hospital organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital Respiratory Medicine, Fukuoka
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Instituto Nacional de Cancerologia, México, D.f., Mexico
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - VUMC, Amsterdam
  - Academisch Ziekenhuis Maastricht / afdeling longziekten en tuberculose, Maastricht
- Oslo universitetssykehus HF - Radiumhospitalet, Oslo, Norway
- Clinica Anglo Americana/Centro de Investigacion Oncologia CAA, San Isidro, Lima region, Peru
- Portugal (4):
  - Centro Hospitalar e Universitario de Coimbra - Hospital Geral, Coimbra
  - Instituto Português de Oncologia de Lisboa, Prof. Francisco Gentil E.P.E., Lisbon
  - Centro Hospitalar de Lisboa Norte - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Russia (6):
  - Russian Oncological Research Center N.N. Blokhin, Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
  - First Saint-Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - First Saint-Petersburg State Medical University n.a. I.P., Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
  - Samara Regional Clinical Oncology Dispensary, Samara
- Singapore (4):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Parkway Cancer Centre, Singapore
  - OncoCare Cancer Centre, Singapore
- South Africa (2):
  - University of Witwatersrand Oncology, Johannesburg, Gauteng
  - Rondebosch Oncology Centre, Rondebosch Medical Centre, Cape Town
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Sungkyunkwan Univ. School of Medicine, Seoul
- Spain (9):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Luzerner Kantonsspital (LUKS), Lucerne
  - Kantonsspital Winterthur, Winterthur
- Taiwan (4):
  - Chang Gung Medical Foundation, Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Comprehensive Cancer Center, Taichung
  - Chang Gung Medical Foundation, LinKou Branch, Taoyuan District
- Ukraine (5):
  - City Multiple-Discipline Clinical Hospital #4,, Dnipropetrovsk
  - City Multiple-Discipline Clinical Hospital #4, Dnipropetrovsk
  - Department of Oncology and Medical Radiology, SI "DMA of MOH, Ukraine, Dnipropetrovsk
  - Kyiv City Clinical Oncologic Center/Department of Chemotherapy, Kyiv
  - Lviv State Oncologic Regional Treatment and Diagnostic Center, Lviv
- United Kingdom (9):
  - Addenbrooke's Hospital, Oncology Centre, Cambridge, Cambridgeshire
  - Lister Hospital, Stevenage, Hertfordshire
  - Queen Elizabeth II Hospital, Welwyn Garden City, Hertfordshire
  - Spire Manchester Hospital, Manchester, Lancashire
  - Mount Vernon Hospital, Mount Vernon Cancer Centre, Northwood, Middlesex
  - NHS Greater Glasgow and Clyde Health Board, Beatson West of Scotland Cancer Centre,, Glasgow, Scotland
  - Ross Hall Hospital, Glasgow, Scotland
  - Aberdeen Royal Infirmary, Aberdeen
  - The Christie Hospital NHS Foundation Trust, Department of Medical Oncology, Manchester

REFERENCES:
- [Derived] Camidge DR, Kim EE, Usari T, Polli A, Lewis I, Wilner KD. Renal Effects of Crizotinib in Patients With ALK-Positive Advanced NSCLC. J Thorac Oncol. 2019 Jun;14(6):1077-1085. doi: 10.1016/j.jtho.2019.02.015. Epub 2019 Feb 26. PMID 30822515
- [Derived] Wilner KD, Usari T, Polli A, Kim EE. Comparison of cardiovascular effects of crizotinib and chemotherapy in ALK-positive advanced non-small-cell lung cancer. Future Oncol. 2019 Apr;15(10):1097-1103. doi: 10.2217/fon-2018-0869. Epub 2019 Jan 17. PMID 30652510
- [Derived] Solomon BJ, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Tang Y, Wilner KD, Blackhall F, Mok TS. Final Overall Survival Analysis From a Study Comparing First-Line Crizotinib Versus Chemotherapy in ALK-Mutation-Positive Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Aug 1;36(22):2251-2258. doi: 10.1200/JCO.2017.77.4794. Epub 2018 May 16. PMID 29768118
- [Derived] Yoneda KY, Scranton JR, Cadogan MA, Tassell V, Nadanaciva S, Wilner KD, Stollenwerk NS. Interstitial Lung Disease Associated With Crizotinib in Patients With Advanced Non-Small Cell Lung Cancer: Independent Review of Four PROFILE Trials. Clin Lung Cancer. 2017 Sep;18(5):472-479. doi: 10.1016/j.cllc.2017.03.004. Epub 2017 Mar 14. PMID 28373069
- [Derived] Solomon BJ, Cappuzzo F, Felip E, Blackhall FH, Costa DB, Kim DW, Nakagawa K, Wu YL, Mekhail T, Paolini J, Tursi J, Usari T, Wilner KD, Selaru P, Mok TS. Intracranial Efficacy of Crizotinib Versus Chemotherapy in Patients With Advanced ALK-Positive Non-Small-Cell Lung Cancer: Results From PROFILE 1014. J Clin Oncol. 2016 Aug 20;34(24):2858-65. doi: 10.1200/JCO.2015.63.5888. Epub 2016 Mar 28. PMID 27022118
- [Derived] Solomon BJ, Mok T, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Iyer S, Reisman A, Wilner KD, Tursi J, Blackhall F; PROFILE 1014 Investigators. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. N Engl J Med. 2014 Dec 4;371(23):2167-77. doi: 10.1056/NEJMoa1408440. PMID 25470694
- [Derived] Ou SH. Crizotinib: a drug that crystallizes a unique molecular subset of non-small-cell lung cancer. Expert Rev Anticancer Ther. 2012 Feb;12(2):151-62. doi: 10.1586/era.11.186. PMID 22316363
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081014&StudyName=A%20Clinical%20Trial%20Testing%20The%20Efficacy%20Of%20Crizotinib%20Versus%20Standard%20Chemotherapy%20Pemetrexed%20Plus%20Cisplatin%20Or%20Carboplatin%20In%20Patients%20With

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with histologically or cytologically proven diagnosis of locally advanced, recurrent, or metastatic non squamous non small cell lung cancer and tumors with measurable disease were enrolled. Participants were to be positive for translocation or inversion events involving the ALK gene locus as determined by an ALK break apart FISH test.
Groups:
- Crizotinib: Crizotinib 250 mg (milligram) capsule, orally twice daily was administered in treatment cycle of 21 days. Participants could continue crizotinib treatment beyond the time of (Response Evaluation Criteria in Solid Tumors) RECIST v1.1 defined PD, as determined by Independent Radiology Review (IRR), at the discretion of the investigator if the participant was perceived to be experiencing clinical benefit.
- Chemotherapy: Standard doses of chemotherapy (pemetrexed/cisplatin or pemetrexed/carboplatin) were administered intravenously on Day 1 of each cycle for a maximum of 6 cycles. Pemetrexed 500 mg per meter square (m)^2 intravenous (IV) infusion according to standard of care was administered over 10 minutes (min); either cisplatin 75 mg/m^2 IV infusion was administered approximately 30 min after the end of the pemetrexed infusion or carboplatin was administered at a dose calculated to produce an area under the concentration time curve (AUC) of 5 or 6 milligram*minute per millilitre (mg*min/mL), approximately 30 min after end of pemetrexed infusion.
Period: Overall Study
Arm/Group | Crizotinib | Chemotherapy
Started | 172 | 171
Treated | 171 | 169
Completed | 81 | 69
Not Completed | 91 | 102
Not completed — Death | 71 | 81
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Other | 3 | 1
Not completed — Randomized but not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis (FA) population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Groups:
- Crizotinib: Crizotinib 250 mg capsule, orally twice daily was administered in treatment cycle of 21 days. Participants could continue crizotinib treatment beyond the time of RECIST v1.1 defined PD, as determined by IRR, at the discretion of the investigator if the participant was perceived to be experiencing clinical benefit.
- Chemotherapy: Standard doses of chemotherapy (pemetrexed/cisplatin or pemetrexed/carboplatin) were administered intravenously on Day 1 of each cycle for a maximum of 6 cycles. Pemetrexed 500 mg per meter square (m)^2 IV infusion according to standard of care was administered over 10 min; either cisplatin 75 mg/m^2 IV infusion was administered approximately 30 min after the end of the pemetrexed infusion or carboplatin was administered at a dose calculated to produce an AUC of 5 or 6 mg*min/mL, approximately 30 min after end of pemetrexed infusion.
- Total: Total of all reporting groups
Arm/Group | Crizotinib | Chemotherapy | Total
Number analyzed (Participants) | 172 | 171 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.94 (11.9) | 52.89 (13.1) | 51.92 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 108 | 212
  Male | 68 | 63 | 131

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on IRR
Description: PFS was defined as the time from the date of randomization in study until the date of first documented objective tumor progression (according to RECIST v1.1 as determined by IRR) or death (due to any cause), whichever occurred first. PFS (in months) was calculated as (first event date - randomization date +1)/30.44. Objective progression was defined as a 20 percent (%) increase in the sum of the diameters of target measurable lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), with a minimum absolute increase of 5 millimeter (mm) or clear progression of pre-existing non-target lesions, or the appearance of any new clear lesions.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression before any additional anti-cancer therapy (up to 35 months)
Population: The FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
months | 10.9 [8.3 to 13.9] | 7.0 [6.8 to 8.2]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value was obtained from 1-sided log rank test, stratified by eastern cooperative oncology group performance status (ECOG PS),race,brain metastases. 1-sided log-rank test at 0.0247 level of significance was used to compare PFS between the 2 arms; Hazard Ratio (HR) = 0.454, 95% CI 2-sided [0.346 to 0.596]

2. Secondary Outcome: Overall Survival (OS)
Description: OS (in months) was defined as the duration from start of study treatment to date of death due to any cause. OS = (date of death minus the date of randomization of study medication plus 1) divided by 30.4. For participants who were alive, overall survival was censored on last date the participants were known to be alive.
Time Frame: From randomization to death or last date known alive for those not known to have died (up to 72 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
months | NA [45.8 to NA] — Median and upper limit of 95% CI were not estimable due to the small number of participants who had event. | 47.5 [32.2 to NA] — Upper limit of 95% CI was not estimable due to the small number of participants who had event.
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p = 0.0489, Log Rank — P-value was obtained from 1-sided log rank test, stratified by ECOG PS, race group and brain metastases; Hazard Ratio (HR) = 0.760, 95% CI 2-sided [0.548 to 1.053] — HR was calculated based on the Cox Proportional hazards model stratified by ECOG PS, race group, and brain metastases. Assuming proportional hazards, a hazard ratio (less than)<1 indicates a reduction in hazard rate in favor of crizotinib

3. Secondary Outcome: Overall Survival Probability at Month 12 and 18
Description: Overall survival probability at Month 12 and 18 was defined as the probability of overall survival at 12 and 18 months respectively, where the OS was defined as the duration from date of randomization to date of death due to any cause. The survival probability was estimated using the Kaplan-Meier method.
Time Frame: Month 12, 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
percent probability
  Month 12 | 83.5 [77.0 to 88.3] | 78.4 [71.3 to 83.9]
  Month 18 | 71.5 [64.0 to 77.7] | 66.6 [58.8 to 73.2]

4. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response as Assessed by IRR
Description: ORR was defined as percentage of participants with complete response (CR) or partial response (PR) according to RECIST v1.1 determined by IRR. CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as greater than or equal to (>=) 30% decrease taking as reference the baseline sum of lesion dimensions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No clear progression of non-target disease. No new lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
percentage of participants | 74.4 [67.2 to 80.8] | 45.0 [37.4 to 52.8]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; If the PFS endpoint was significant, ORR was to be considered significant if the 2-sided p-value from Pearson chi-square test was (less than or equal to)<= 0.0494; Test type: Superiority or Other; p < 0.0001, Pearson chi-square test — P-value was obtained from a Pearson chi-square test; Difference in Percentage = 29.4, 95% CI 2-sided [19.5 to 39.3] — 95% CI was calculated based on normal distribution

5. Secondary Outcome: Duration of Response (DR) Based on IRR
Description: DR: time from first documentation of objective tumor response (CR or PR) to first documentation of PD or death due to any cause, whichever occurred first as per RECIST v1.1 determined by IRR. CR: complete disappearance of all target and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions, disappearance of all non-target lesions. PR: >=30% decrease taking as reference the baseline sum of lesion dimensions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all or target lesions. No clear progression of non-target disease. No new lesions. c) PD: 20 % increase in the sum of the diameters of target measurable lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), with a minimum absolute increase of 5 mm or clear progression of pre-existing non-target lesions, or the appearance of any new clear lesions.
Time Frame: From objective response to date of progression, death or last tumor assessment without progression before any additional anti-cancer therapy (up to 35 months)
Population: The FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization. Here Overall number of participants analyzed (N) signifies participants with objective tumor response and were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 128 | 77
weeks | 49.0 [35.1 to 60.0] | 22.9 [18.0 to 25.1]

6. Secondary Outcome: Time to Tumor Response (TTR) Based on IRR
Description: TTR was defined as the time from randomization to first documentation of objective tumor response (CR or PR) according to RECIST v1.1 determined by IRR. CR: complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR: >=30% decrease taking as reference the baseline sum of lesion dimensions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all or target lesions. No clear progression of non-target disease. No new lesions.
Time Frame: Randomization to first documentation of objective tumor response (up to 35 months)
Population: The FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization. Here N signifies participants with objective tumor response and were evaluable for this outcome measure.
Measure: Median (Full Range); unit: weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 128 | 77
weeks | 6.1 [2.7 to 41.4] | 12.1 [5.1 to 36.7]

7. Secondary Outcome: Percentage of Participants With Disease Control at Week 12 Based on IRR
Description: Disease control rate at week 12 is defined as the percent of participants with CR, PR, or stable disease (SD) at week 12 according to RECIST v1.1 determined by IRR. The best response of SD would be assigned if SD criteria was met at least once after randomization at a minimum interval of 6 weeks. CR: complete disappearance of all target lesions and non-target disease, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR: >=30% decrease taking as reference the baseline sum of lesion dimensions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters. Short axis was used in sum for target nodes, while longest diameter was used in sum for all or target lesions. No clear progression of non-target disease. No new lesions.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
percentage of participants | 78.5 [71.6 to 84.4] | 68.4 [60.9 to 75.3]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; The confidence interval for the difference in percentage was based on normal distribution; Test type: Superiority or Other; p = 0.0381, Pearson chi-square test; Difference in Percentage = 10.067, 95% CI 2-sided [0.8 to 19.4]

8. Secondary Outcome: Time to Progression (TTP) Based on IRR
Description: TTP was defined as the time from the date of randomization to the date of the first documentation of objective tumor progression according to RECIST v1.1 determined by IRR. Objective tumor progression was defined as 20% increase in the sum of the diameters of target measurable lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), with a minimum absolute increase of 5 mm or clear progression of pre-existing non-target lesions, or the appearance of any new clear lesions. If tumor progression data included more than 1 date, the first date was used. TTP (in months) was calculated as (first event date - randomization date +1)/30.44.
Time Frame: Randomization to objective progression or last tumor assessment without progression before any additional anti-cancer therapy (up to 35 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
months | 13.6 [8.5 to 15.0] | 7.0 [6.8 to 8.3]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis was based on the Cox Proportional hazards model assuming proportional hazards, a HR <1 indicated a reduction in hazard rate in favor of Crizotinib; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value was obtained from 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.441, 95% CI 2-sided [0.335 to 0.582]

9. Secondary Outcome: Time to Intracranial Progression (IC-TTP) Based on IRR
Description: IC-TTP was defined similarly to TTP, but only considering intracranial disease (excluding extracranial disease) and the progression was determined based on either new brain metastases or progression of existing brain metastases. TTP was defined as the time from the date of randomization to the date of the first documentation of objective tumor progression according to RECIST v1.1 determined by IRR. Objective tumor progression was defined as 20% increase in the sum of the diameters of target measurable lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), with a minimum absolute increase of 5 mm or clear progression of pre-existing non-target lesions, or the appearance of any new clear lesions.
Time Frame: Randomization to objective intracranial progression or last tumor assessment without progression before any additional anti-cancer therapy (up to 35 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
months | NA [NA to NA] — Median and CI were not reached due to immaturity of data and low number of events. | 17.8 [13.9 to NA] — Upper limit of 95% CI was not estimable due to the small number of participants who had event.
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis was based on the Cox Proportional hazards model assuming proportional hazards, a HR less than 1 indicated a reduction in hazard rate in favor of Crizotinib; Test type: Superiority or Other; p = 0.0347, Log Rank — P-value was obtained from 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.595, 95% CI 2-sided [0.338 to 1.048]

10. Secondary Outcome: Time to Extracranial Progression (EC-TTP) Based on IRR
Description: EC-TTP was defined similarly to TTP, but only considering extracranial disease (excluding intracranial disease) and the progression was determined based on either new extracranial lesions or progression of existing extracranial lesions. TTP was defined as the time from the date of randomization to the date of the first documentation of objective tumor progression according to RECIST v1.1 determined by IRR. Objective tumor progression was defined as 20% increase in the sum of the diameters of target measurable lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), with a minimum absolute increase of 5 mm or clear progression of pre-existing non-target lesions, or the appearance of any new clear lesions.
Time Frame: Randomization to objective extracranial progression or last tumor assessment without progression before any additional anti-cancer therapy (up to 35 months)
Population: FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
months | 15.2 [12.6 to 21.9] | 7.2 [6.9 to 8.5]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value was obtained from 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.387, 95% CI 2-sided [0.286 to 0.524]

11. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose of study drug that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: The safety analysis population included all randomized participants who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received during the first cycle.
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 171 | 169
percentage of participants
  AEs | 99.4 | 99.4
  SAEs | 41.5 | 29.0

12. Secondary Outcome: Percentage of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: The safety analysis population included all randomized subjects who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received during the first cycle.
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 171 | 169
percentage of participants
  AEs | 98.2 | 92.3
  SAEs | 12.9 | 8.9

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) According to Maximum Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to maximum severity grading based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Grade 1 =mild; Grade 2 =moderate; within normal limits, Grade 3 =severe or medically significant but not immediately life-threatening; Grade 4 =life-threatening or disabling; urgent intervention indicated; Grade 5 =death.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 171 | 169
percentage of participants
  Grade 1 | 7.0 | 9.5
  Grade 2 | 28.7 | 34.3
  Grade 3 | 41.5 | 44.4
  Grade 4 | 8.8 | 8.9
  Grade 5 | 13.5 | 2.4

14. Secondary Outcome: Plasma Predose Concentration (Ctrough) of Crizotinib and Its Metabolite PF-06260182
Description: Ctrough is the concentration prior to study drug administration on Day 1 of Cycle 2 onwards. PF-06260182 is the metabolite of Crizotinib.
Time Frame: Predose at Day 1 of Cycle 2, 3 and 5
Population: Pharmacokinetic concentration population included all participants in the safety analysis population who had at least 1 plasma concentration of crizotinib or its metabolite.N=participants evaluable for this measure.Number of participants analyzed(n)=participants evaluable at specified time points.This analysis was performed in crizotinib arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Crizotinib
Number analyzed (Participants) | 162
nanogram per milliliter
  Crizotinib Ctrough: Cycle 2 Day 1: number analyzed (Participants) | 91
  Crizotinib Ctrough: Cycle 2 Day 1 | 324.2 (39)
  Crizotinib Ctrough: Cycle 3 Day 1: number analyzed (Participants) | 85
  Crizotinib Ctrough: Cycle 3 Day 1 | 320.9 (40)
  Crizotinib Ctrough: Cycle 5 Day 1: number analyzed (Participants) | 82
  Crizotinib Ctrough: Cycle 5 Day 1 | 308.2 (39)
  PF-06260182 Ctrough: Cycle 2 Day 1: number analyzed (Participants) | 100
  PF-06260182 Ctrough: Cycle 2 Day 1 | 98.4 (46)
  PF-06260182 Ctrough: Cycle 3 Day 1: number analyzed (Participants) | 94
  PF-06260182 Ctrough: Cycle 3 Day 1 | 99.0 (49)
  PF-06260182 Ctrough: Cycle 5 Day 1: number analyzed (Participants) | 86
  PF-06260182 Ctrough: Cycle 5 Day 1 | 92.9 (55)

15. Secondary Outcome: Percentage of Participants For Each Anaplastic Lymphoma Kinase (ALK) Gene Fusion Variants
Description: The Response Genetics, Inc. Echinoderm Microtubule Associated Protein Like 4 (EML4) ALK reverse transcriptase polymerase chain reaction (RT PCR) gene fusion test was used for the analysis of tissue samples for the ALK gene fusion variants (either no rearrangement, or 1 of 9 results reflecting 8 specific rearrangements [V1, V2, V3a, V3b,V3a/b, V4, V5a, V6, V7]). Percentage of participants who tested positive for ALK gene fusion variants were reported in this outcome measure.
Time Frame: 28 days prior to day 1 of study treatment
Population: The ALK variant evaluable population included participants from the FA population who had a result from ALK gene fusion variant testing of either no rearrangement, or 1 of 9 results reflecting 8 specific rearrangements (V1, V2, V3a, V3b, V3a/b, V4, V5a, V6, and V7).
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 70 | 78
percentage of participants
  V1 | 27.1 | 25.6
  V2 | 7.1 | 7.7
  V3a | 1.4 | 1.3
  V3a/b | 4.3 | 6.4
  No rearrangement | 60.0 | 59.0

16. Secondary Outcome: Objective Response Rate (ORR) of Anaplastic Lymphoma Kinase (ALK) Variant Groups Based on IRR
Description: The Response Genetics, Inc. EML4 ALK reverse transcriptase polymerase chain reaction (RT PCR) gene fusion test was used for the analysis of tissue samples for the ALK gene fusion variants (either no rearrangement, or 1 of 9 results reflecting 8 specific rearrangements [V1, V2, V3a, V3b,V3a/b, V4, V5a, V6, V7]). Percentage of participants with confirmed CR or PR according to RECIST v1.1 determined by IRR, by type of ALK gene fusion variant were reported in this outcome measure. CR: complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR: >=30% decrease decrease taking as reference the baseline sum of lesion dimensions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all or target lesions. No clear progression of non-target disease. No new lesions.
Time Frame: as for outcome 1
Population: The ALK variant evaluable population included participants from the FA population who had a result from ALK gene fusion variant testing of either no rearrangement, or 1 of 9 results reflecting 8 specific rearrangements (V1, V2, V3a, V3b, V3a/b, V4, V5a, V6, and V7). Here, n signifies participants who were evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 70 | 78
percentage of participants
  V1: number analyzed (Participants) | 19 | 20
  V1 | 84.2 [60.4 to 96.6] | 45.0 [23.1 to 68.5]
  V2: number analyzed (Participants) | 5 | 6
  V2 | 100 [47.8 to 100] | 33.3 [4.3 to 77.7]
  V3a: number analyzed (Participants) | 1 | 1
  V3a | 0.0 [NA to NA] — Upper and lower limit of 95% CI was not estimable as the percentage of participants were 0.0 for this specific strain. | 100 [2.5 to 100]
  V3a/b: number analyzed (Participants) | 3 | 5
  V3a/b | 100 [29.2 to 100] | 60.0 [14.7 to 94.7]
  No rearrangement: number analyzed (Participants) | 42 | 46
  No rearrangement | 71.4 [55.4 to 84.3] | 43.5 [28.9 to 58.9]

17. Secondary Outcome: Time to Deterioration (TTD) in Chest Pain, Dyspnea or Cough
Description: TTD in pain in chest, dyspnea, or cough from the Quality of Life Questionnaire Core 30 (QLQ-LC13) was a composite endpoint defined as the time from randomization to the earliest time the participant's scale scores showed a 10 point or greater increase after baseline in any of the 3 symptoms. For those who had not shown deterioration, the data was censored at the last date when the participants completed an assessment (QLQ-LC13) for pain, dyspnea, or cough or at last visit date prior to crossover for participants randomized to chemotherapy who subsequently crossed over to crizotinib. A 10-point or higher change in the score was perceived by participants as clinically significant. The transformed score of pain, dyspnea, and cough symptom scales of EORTC QLQ-LC13 (European Organization for the Research and Treatment of Cancer) range from 0 to 100, where higher scores indicate greater symptom severity.
Time Frame: From randomization of treatment up to deterioration while on study treatment (up to 35 months)
Population: The patient reported outcome (PRO) evaluable population included all participants from the FA population who completed a baseline and at least 1 postbaseline PRO assessment prior to crossover to crizotinib or end of randomized study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 166 | 163
months | 2.1 [0.8 to 4.2] | 0.5 [0.4 to 0.7]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; HR was calculated based on the Cox Proportional hazards model. Assuming proportional hazards, a HR less than 1 indicated a reduction in hazard rate in favor of crizotinib; Test type: Superiority or Other; p = 0.0002, Log Rank — Two-sided p-value from the unstratified log rank test was used; Hazard Ratio (HR) = 0.591, 95% CI 2-sided [0.452 to 0.773]

18. Secondary Outcome: Change From Baseline in Functioning and Global Quality of Life (QOL) as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: EORTC QLQ-C30: included 5 functional scales (physical, role, cognitive, emotional and social), global health status/global quality of life scale, 3 symptom scales (fatigue, pain, nausea and vomiting), 6 single items that assess the additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, diarrhea) and financial difficulties. All scales and single-item measures range from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, for the global health status/QoL represents a high QoL (better participant state), and for a symptom scale/item represents a high level of symptoms/problems (worse participant state).
Time Frame: Baseline, From Cycle 1 Day 1 up to end of study treatment or crossover to crizotinib arm (up to 35 months)
Population: The PRO evaluable population included all participants from the FA population who completed a baseline and at least 1 postbaseline PRO assessment prior to crossover to crizotinib or end of randomized study treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 166 | 163
units on a scale
  QLQ-C30 Global QoL | 5.9815 [3.92 to 8.05] | -7.8488 [-10.15 to -5.55]
  QLQ-C30 Cognitive Functioning | 1.1836 [-0.66 to 3.03] | -2.1696 [-4.21 to -0.13]
  QLQ-C30 Emotional Functioning | 8.7431 [6.77 to 10.72] | 1.2266 [-0.95 to 3.40]
  QLQ-C30 Physical Functioning | 5.9370 [3.94 to 7.93] | -4.4664 [-6.59 to -2.34]
  QLQ-C30 Role Functioning | 4.8122 [1.92 to 7.71] | -10.7391 [-13.87 to -7.61]
  QLQ-C30 Social Functioning | 4.3790 [1.60 to 7.15] | -4.3851 [-7.37 to -1.40]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 Global QoL: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 13.8303, 95% CI 2-sided [10.74 to 16.92]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 cognitive functioning: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0170, Mixed Models Analysis; Mean Difference (Net) = 3.3532, 95% CI 2-sided [0.60 to 6.11]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 emotional functioning: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 7.5165, 95% CI 2-sided [4.57 to 10.46]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 physical functioning: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 10.4035, 95% CI 2-sided [7.48 to 13.32]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 role functioning: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 15.5513, 95% CI 2-sided [11.29 to 19.81]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 social functioning: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 8.7641, 95% CI 2-sided [4.69 to 12.84]

19. Secondary Outcome: Change From Baseline Scores in QLQ-C30 Symptoms as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: as for outcome 18
Time Frame: Baseline, From Cycle 1 Day 1 up to end of study treatment or crossover to crizotinib arm (up to 35 months)
Population: as for outcome 18
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 166 | 163
units on a scale
  QLQ-C30 Appetite loss | -5.4906 [-8.52 to -2.47] | 8.0070 [4.63 to 11.38]
  QLQ-C30 Constipation | 6.4858 [3.46 to 9.51] | 10.9194 [7.50 to 14.34]
  QLQ-C30 Diarrhea | 12.9558 [10.67 to 15.24] | 0.4652 [-2.20 to 3.13]
  QLQ-C30 Dysponea | -14.9019 [-17.40 to -12.40] | -1.4398 [-4.21 to 1.33]
  QLQ-C30 Fatigue | -7.3476 [-9.72 to -4.98] | 7.6511 [5.05 to 10.25]
  QLQ-C30 Financial Difficulties | -0.5984 [-3.13 to 1.93] | 0.2203 [-2.54 to 2.98]
  QLQ-C30 Insomnia | -10.3095 [-13.10 to -7.52] | -0.2665 [-3.38 to 2.84]
  QLQ-C30 Nausea and Vomiting | 3.7742 [1.54 to 6.01] | 7.2188 [4.66 to 9.78]
  QLQ-C30 Pain | -11.0993 [-13.27 to -8.92] | -1.1716 [-3.66 to 1.31]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 appetite loss: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -13.4976, 95% CI 2-sided [-18.03 to -8.97]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 constipation: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0570, Mixed Models Analysis; Mean Difference (Net) = -4.4336, 95% CI 2-sided [-9.00 to 0.13]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 diarrhea: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 12.4906, 95% CI 2-sided [8.98 to 16.00]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 dysponea: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Median Difference (Net) = -13.4622, 95% CI 2-sided [-17.20 to -9.73]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 fatigue: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -14.9987, 95% CI 2-sided [-18.52 to -11.48]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 financial difficulties: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.6681, Mixed Models Analysis; Mean Difference (Net) = -0.8186, 95% CI 2-sided [-4.56 to 2.92]
Statistical Analysis 7: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 insomnia: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -10.0430, 95% CI 2-sided [-14.22 to -5.87]
Statistical Analysis 8: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 nausea and vomiting: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0468, Mixed Models Analysis; Mean Difference (Net) = -3.4446, 95% CI 2-sided [-6.84 to -0.05]
Statistical Analysis 9: Comparison: Crizotinib vs Chemotherapy; QLQ-C30 pain: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -9.9277, 95% CI 2-sided [-13.23 to -6.62]

20. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scores as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 (QLQ- LC13)
Description: QLQ-LC13 consists of 1 multi-item scale and 9 single items that assess the specific symptoms (dyspnea, cough, hemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of patients with lung cancer receiving chemotherapy. All multi-item scales and single-item measures range from 0 to 100, where higher score indicates greater degree of symptom severity.
Time Frame: Baseline, From Cycle 1 Day 1 up to end of study treatment or crossover to crizotinib arm (up to 35 months)
Population: as for outcome 18
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 166 | 163
units on a scale
  QLQ-LC13 Alopecia | -4.4879 [-6.99 to -1.99] | 0.3271 [-2.40 to 3.06]
  QLQ-LC13 Coughing | -16.4819 [-18.92 to -14.05] | -8.0893 [-10.83 to -5.35]
  QLQ-LC13 Dysphagia | 0.7618 [-0.82 to 2.35] | 0.09660 [-1.76 to 1.95]
  QLQ-LC13 Dyspnoea | -9.2029 [-11.20 to -7.20] | -0.1948 [-2.36 to 1.97]
  QLQ-LC13 Haemoptysis | -3.2197 [-3.83 to -2.61] | -2.3369 [-3.05 to -1.62]
  QLQ-LC13 Pain in Arm or Shoulder | -10.1693 [-12.26 to -8.08] | -4.1218 [-6.51 to -1.74]
  QLQ-LC13 Pain in Chest | -8.1437 [-10.31 to -5.98] | -0.04790 [-2.48 to 2.38]
  QLQ-LC13 Pain in Other Parts | -8.0757 [-10.28 to -5.87] | -1.3040 [-3.97 to 1.36]
  QLQ-LC13 Peripheral Neuropathy | 3.1779 [1.04 to 5.31] | -0.1742 [-2.60 to 2.25]
  QLQ-LC13 Sore Mouth | 2.2472 [0.36 to 4.13] | 4.3993 [2.27 to 6.53]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 alopecia: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0108, Mixed Models Analysis; Mean Difference (Net) = -4.8149, 95% CI 2-sided [-8.52 to -1.11]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 coughing: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -8.3926, 95% CI 2-sided [-12.06 to -4.72]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 dysphagia: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.5938, Mixed Models Analysis; Mean Difference (Net) = 0.6651, 95% CI 2-sided [-1.78 to 3.11]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 dyspnoea: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -9.0080, 95% CI 2-sided [-11.96 to -6.06]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 haemoptysis: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0656, Mixed Models Analysis; Mean Difference (Net) = -0.8828, 95% CI 2-sided [-1.82 to 0.06]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 pain in arm or shoulder: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -6.0475, 95% CI 2-sided [-9.22 to -2.88]
Statistical Analysis 7: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 pain in chest: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -8.0959, 95% CI 2-sided [-11.35 to -4.84]
Statistical Analysis 8: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 pain in other parts: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Net) = -6.7717, 95% CI 2-sided [-10.24 to -3.31]
Statistical Analysis 9: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 peripheral neuropathy: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.0427, Mixed Models Analysis; Mean Difference (Net) = 3.3521, 95% CI 2-sided [0.11 to 6.59]
Statistical Analysis 10: Comparison: Crizotinib vs Chemotherapy; QLQ-LC13 sore mouth: Analysis was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects); Test type: Superiority or Other; p = 0.1382, Mixed Models Analysis; Mean Difference (Net) = -2.1521, 95% CI 2-sided [-5.00 to 0.69]

21. Secondary Outcome: Change From Baseline in General Health Status as Assessed by EuroQol 5D (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. VAS component: participants rated their current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health.
Time Frame: Baseline, From Cycle 1 Day 1 up to end of study treatment or crossover to crizotinib arm (up to 35 months)
Population: The patient reported outcome (PRO) evaluable population included all participants from the FA population who completed a baseline and at least 1 postbaseline PRO assessment prior to crossover to crizotinib or end of randomized study treatment. Here, "N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 160 | 160
units on a scale | 4.5323 [2.44 to 6.62] | 0.5415 [-1.85 to 2.93]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis was based on a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EQ-5D VAS subscale baseline score (intercept and time from first dose were included as random effects); Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; Mean Difference (Net) = 3.9908, 95% CI 2-sided [0.81 to 7.17]

22. Secondary Outcome: Percentage of Participants With Hospital Admissions-Healthcare Resource Utilization (HCRU)
Description: Healthcare resource utilization was to be evaluated using the assessment of the following: date and duration of index admission, duration of hospitalization and date of discharge.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 172 | 171
percentage of participants | 40.12 | 36.26

23. Secondary Outcome: Percentage of Participants With Laboratory Test Abnormalities By Maximum Severity: National Cancer Institute Common Terminology Criteria for Adverse Event (Version 4.0) Grade 1 to 4 Hematological Test Abnormalities
Description: Anemia(grade[g]1:Less than[<] Lower limit of normal[LLN] to 10gram per[/] deciliter[g/dL],g2:<10 to 8g/dL,g3:<8g/dL,g4:lifethreatening);platelet (g1:<LLN to 75*10^3/millimeter[mm]^3,g2:<75*10^3/mm^3 to 50*10^3/mm^3,g3:<50*10^3/mm^3 to 25*10^3/mm^3,g4:<25*10^3/mm^3);lymphopenia(g1:<LLN to 8*10^2/mm^3,g2:<8*10^2 to 5*10^2/mm^3,g3:<5*10^2 to 2*10^2/mm^3,g4:<2*10^2/mm^3);neutrophil (Absolute)(g1:<LLN to 15*10^2/mm^3,g2:<15*10^2 to 10*10^2/mm^3,g3:<10*10^2 to 5*10^2/mm^3,g4:<5*10^2/mm^3);white blood cell count(g1:<LLN to 3*10^3/mm^3,g2:<3*10^3 to 2*10^3/mm^3,g3:<2*10^3 to 1*10^3/mm^3,g4:<1*10^3/mm^3);hemoglobin(g1:increase in hemoglobin level>0 to 2 g/dL above ULN or above baseline if baseline is above ULN,g2:increase in hemoglobin level>2 to 4g/dL above ULN or above baseline if baseline is above ULN,g3:increase in hemoglobin level>4 g/dL above ULN or above baseline if baseline is above ULN). Only categories with atleast 1 participant with abnormality are reported in this outcome measure.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: Safety analysis population included all randomized subjects who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received during the first cycle. Here, N=participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 170 | 165
percentage of participants
  Anemia: Grade 1 | 47.1 | 46.7
  Anemia: Grade 2 | 13.5 | 27.9
  Anemia: Grade 3 | 0.6 | 10.9
  Hemoglobin increased: Grade 1 | 6.5 | 3.0
  Hemoglobin increased: Grade 2 | 0.6 | 0.0
  Lymphocyte count increased: Grade 2 | 3.5 | 1.2
  Lymphopenia: Grade 1 | 34.1 | 26.1
  Lymphopenia: Grade 2 | 24.7 | 33.9
  Lymphopenia: Grade 3 | 10.6 | 13.9
  Lymphopenia: Grade 4 | 2.4 | 1.8
  Neutrophils (Absolute): Grade 1 | 20.6 | 14.5
  Neutrophils (Absolute): Grade 2 | 20.0 | 26.7
  Neutrophils (Absolute): Grade 3 | 14.1 | 13.9
  Neutrophils (Absolute): Grade 4 | 0.6 | 3.6
  Platelets: Grade 1 | 9.4 | 21.8
  Platelets: Grade 2 | 2.4 | 7.9
  Platelets: Grade 3 | 0.6 | 7.9
  Platelets: Grade 4 | 0.0 | 0.6
  White blood cells: Grade 1 | 23.5 | 34.5
  White blood cells: Grade 2 | 22.9 | 24.2
  White blood cells: Grade 3 | 2.9 | 9.1
  White blood cells: Grade 4 | 0.0 | 0.6

24. Secondary Outcome: Percentage of Participants With Laboratory Test Abnormalities By Maximum Severity: National Cancer Institute Common Terminology Criteria for Adverse Event (Version 4.0) Grade 1 to 4 Chemistry Test Abnormalities
Description: ALT/AST (Grade[g]1:>ULN-3*ULN,g2:>3-5*ULN,g3:>5-20*ULN,g4:>20*ULN);Alkaline Phosphatase (g1:>ULN-2.5*ULN,g2:>2.5-5*ULN,g3:>5-20*ULN,g4:>20*ULN);Creatinine (g1:>ULN-1.5*ULN,g2:>1.5-3*ULN,g3:>3-6*ULN,g4:>6*ULN);hyperglycemia (g1:>ULN-160,g2:>160-250,g3:>250-500,g4:>500mg/dL);bilirubin(total) (g1:>ULN-1.5*ULN,g2:>1.5-3*ULN,g3:>3-10*ULN,g4:>10*ULN);hypoglycaemia (g1:<LLN-55,g2:<55-40,g3:<40-30,g4:<30mg/dL);hyperkalemia (g1:>ULN-5.5,g2:>5.5-6,g3:>6-7,g4:>7mmol/L);hypokalemia (g1:<LLN-3,g2:<LLN-3,g3:<3-2.5,g4:<2.5mmol/L);hypermagnesemia (g1:>ULN-3,g3:>3-8,g4:>8mg/dL);hypocalcemia (g1:<LLN-8,g2:<8-7,g3:<7-6,g4:<6mg/dL); hypercalcemia (g1:>ULN-11.5,g2:>11.5-12.5,g3:>12.5-13.5,g4:>13.5mg/dL);hypomagnesemia (g1:<LLN-1.2,g2:<1.2-0.9,g3:<0.9-0.7,g4:<0.7mg/dL);hyponatremia (g1:<LLN-130,g3:<130-120,g4:<120mmol/L);hypoalbuminemia (g1:<LLN-3,g2:<3-2,g3:<2,g4:lifethreatening);hypophosphatemia (g1:<LLN-2.5,g2:<2.5-2,g3:<2-1,g4:<1mg/dL). Participant>=1 abnormality given.
Time Frame: Baseline up to follow up period (up to 72 months)
Population: Safety analysis population included all randomized subjects who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received during the first cycle. Here, N=participants who were evaluable for this outcome measure. Here, "n"=participants who were evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 171 | 165
percentage of participants
  Alanine aminotransferase: Grade 1 | 64.3 | 34.5
  Alanine aminotransferase: Grade 2 | 10.5 | 7.3
  Alanine aminotransferase: Grade 3 | 12.3 | 1.8
  Alanine aminotransferase: Grade 4 | 2.3 | 0.0
  Alkaline phosphatase: Grade 1 | 55.6 | 33.9
  Alkaline phosphatase: Grade 2 | 8.8 | 4.8
  Alkaline phosphatase: Grade 3 | 0.6 | 1.2
  Aspartate Aminotransferase: Grade 1 | 57.9 | 32.1
  Aspartate Aminotransferase: Grade 2 | 6.4 | 1.8
  Aspartate Aminotransferase: Grade 3 | 7.6 | 1.2
  Aspartate Aminotransferase: Grade 4 | 0.6 | 0.0
  Bilirubin: Grade 1 | 10.5 | 7.3
  Bilirubin: Grade 2 | 5.8 | 1.2
  Bilirubin: Grade 3 | 0.0 | 0.6
  Creatinine: Grade 1 | 50.3 | 78.8
  Creatinine: Grade 2 | 47.4 | 15.8
  Creatinine: Grade 3 | 1.2 | 0.0
  Hypercalcemia: Grade 1 | 0.6 | 9.1
  Hypercalcemia: Grade 4 | 0.6 | 0.0
  Hyperglycemia: Grade 1 | 50.3 | 42.4
  Hyperglycemia: Grade 2 | 15.8 | 23.6
  Hyperglycemia: Grade 3 | 4.1 | 3.6
  Hyperkalemia: Grade 1 | 17.5 | 12.1
  Hyperkalemia: Grade 2 | 5.8 | 3.0
  Hyperkalemia: Grade 3 | 2.3 | 1.8
  Hyperkalemia: Grade 4 | 0.6 | 0.0
  Hypermagnesemia: Grade 1: number analyzed (Participants) | 171 | 162
  Hypermagnesemia: Grade 1 | 17.6 | 8.0
  Hypermagnesemia: Grade 3: number analyzed (Participants) | 171 | 162
  Hypermagnesemia: Grade 3 | 1.8 | 0.0
  Hypernatremia: Grade 1 | 21.1 | 5.5
  Hypernatremia: Grade 2 | 0.6 | 0.0
  Hypernatremia: Grade 4 | 0.6 | 0.0
  Hypoalbuminemia: Grade 1: number analyzed (Participants) | 171 | 164
  Hypoalbuminemia: Grade 1 | 35.1 | 22.6
  Hypoalbuminemia: Grade 2: number analyzed (Participants) | 171 | 164
  Hypoalbuminemia: Grade 2 | 44.4 | 14.6
  Hypoalbuminemia: Grade 3: number analyzed (Participants) | 171 | 164
  Hypoalbuminemia: Grade 3 | 1.2 | 0.6
  Hypocalcemia: Grade 1 | 39.8 | 24.8
  Hypocalcemia: Grade 2 | 38.0 | 4.8
  Hypocalcemia: Grade 3 | 2.3 | 0.6
  Hypoglycemia: Grade 1 | 19.9 | 3.6
  Hypoglycemia: Grade 2 | 4.7 | 1.8
  Hypoglycemia: Grade 4 | 0.0 | 0.6
  Hypokalemia: Grade 1 | 14.6 | 9.1
  Hypokalemia: Grade 3 | 2.3 | 3.0
  Hypokalemia: Grade 4 | 0.0 | 0.6
  Hypomagnesemia: Grade 1 (n =170, 162): number analyzed (Participants) | 170 | 162
  Hypomagnesemia: Grade 1 (n =170, 162) | 12.4 | 26.5
  Hypomagnesemia: Grade 2: number analyzed (Participants) | 170 | 162
  Hypomagnesemia: Grade 2 | 0.0 | 1.9
  Hyponatremia: Grade 1 | 25.7 | 22.4
  Hyponatremia: Grade 3 | 4.1 | 5.5
  Hyponatremia: Grade 4 | 0.6 | 1.2
  Hypophosphatemia: Grade 1: number analyzed (Participants) | 169 | 161
  Hypophosphatemia: Grade 1 | 5.3 | 3.1
  Hypophosphatemia: Grade 2: number analyzed (Participants) | 169 | 161
  Hypophosphatemia: Grade 2 | 27.2 | 13.0
  Hypophosphatemia: Grade 3: number analyzed (Participants) | 169 | 161
  Hypophosphatemia: Grade 3 | 13.0 | 6.8
  Hypophosphatemia: Grade 4: number analyzed (Participants) | 169 | 161
  Hypophosphatemia: Grade 4 | 1.2 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline up to follow up period (up to 72 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 71/171 | 49/169
Other Adverse Events (participants affected / at risk) | 169/171 | 164/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Crizotinib (N=171) | Chemotherapy (N=169)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Syncope (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4
Chest pain (General disorders) | 1 | 1
Disease progression (General disorders) | 18 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Hypomania (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 5
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/104 | 0/108 — This adverse event is gender specific.
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1/104 | 0/108 — This adverse event is gender specific.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=171) | Chemotherapy (N=169)
Anaemia (Blood and lymphatic system disorders) | 18 | 53
Leukopenia (Blood and lymphatic system disorders) | 8 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 14
Bradycardia (Cardiac disorders) | 22 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 10
Photopsia (Eye disorders) | 18 | 2
Vision blurred (Eye disorders) | 13 | 5
Visual impairment (Eye disorders) | 98 | 5
Vitreous floaters (Eye disorders) | 11 | 1
Abdominal pain (Gastrointestinal disorders) | 25 | 8
Abdominal pain upper (Gastrointestinal disorders) | 27 | 10
Constipation (Gastrointestinal disorders) | 78 | 51
Diarrhoea (Gastrointestinal disorders) | 111 | 22
Dyspepsia (Gastrointestinal disorders) | 27 | 5
Dysphagia (Gastrointestinal disorders) | 19 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 6
Nausea (Gastrointestinal disorders) | 100 | 98
Stomatitis (Gastrointestinal disorders) | 13 | 17
Vomiting (Gastrointestinal disorders) | 87 | 57
Asthenia (General disorders) | 28 | 40
Chest pain (General disorders) | 21 | 14
Fatigue (General disorders) | 54 | 66
Mucosal inflammation (General disorders) | 2 | 9
Oedema peripheral (General disorders) | 89 | 12
Pyrexia (General disorders) | 40 | 17
Nasopharyngitis (Infections and infestations) | 30 | 5
Upper respiratory tract infection (Infections and infestations) | 41 | 13
Alanine aminotransferase increased (Investigations) | 59 | 21
Aspartate aminotransferase increased (Investigations) | 47 | 16
Electrocardiogram QT prolonged (Investigations) | 11 | 2
Neutrophil count decreased (Investigations) | 14 | 17
Platelet count decreased (Investigations) | 1 | 19
Weight decreased (Investigations) | 12 | 5
Weight increased (Investigations) | 16 | 4
White blood cell count decreased (Investigations) | 11 | 12
Decreased appetite (Metabolism and nutrition disorders) | 59 | 58
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 14
Dizziness (Nervous system disorders) | 35 | 15
Dysgeusia (Nervous system disorders) | 45 | 9
Headache (Nervous system disorders) | 48 | 25
Neuropathy peripheral (Nervous system disorders) | 4 | 12
Paraesthesia (Nervous system disorders) | 29 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 10
Anxiety (Psychiatric disorders) | 10 | 9
Insomnia (Psychiatric disorders) | 23 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 10
Rash (Skin and subcutaneous tissue disorders) | 22 | 20
Neutropenia (Blood and lymphatic system disorders) | 32 | 36
Sinus bradycardia (Cardiac disorders) | 10 | 1
Abdominal distension (Gastrointestinal disorders) | 11 | 1
Influenza like illness (General disorders) | 10 | 1
Pain (General disorders) | 9 | 5
Bronchitis (Infections and infestations) | 11 | 2
Conjunctivitis (Infections and infestations) | 3 | 10
Rhinitis (Infections and infestations) | 9 | 2
Urinary tract infection (Infections and infestations) | 10 | 2
Blood bilirubin increased (Investigations) | 9 | 2
Blood creatinine increased (Investigations) | 9 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.